CLINICAL TRIAL: NCT04063241
Title: Parent Understanding of Discharge Instructions
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: After initially being suspended in the setting of the COVID-19 pandemic, the study was then terminated due to lack of funding and staffing to complete it.
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Health Services Research
Other Study IDs: 15-00072
Record Dates: First submitted 2019-08-19; First posted 2019-08-21 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Parent-Child Relations
Keywords: health literacy

STUDY DESIGN:
Intervention Model Description: Parents:
  Phase A (Pre-implementation): Parents in the pre-implementation group will receive standard care: verbal counseling by the doctor/nurse using text-based instructions they have prepared (not standardized). Phase A was completed as an observational study.
  Phase B (Implementation): Provider training (see below) Phase C (Post-implementation): Doctors and nurses will customize the web-based disease-specific instructions with the research team's help. They will reference these instructions as they perform discharge counseling and will give parents a copy of the instructions.
  Providers:
  Pediatric residents knowledge, attitudes, and practices will be assessed at baseline. They will then take part in a 20-minute training session, including information about health literacy, advanced counseling strategies, results of prior studies, and pre-implementation data. Assessments will be performed for those who use the health literacy-informed tool at least once during the study period.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Parent: Pre-implementation (No Intervention): Parents in the pre-implementation group will receive standard care: verbal counseling by the doctor/nurse using text-based instructions they have prepared (not standardized).
- Parent: Post-Implementation (Experimental): Doctors and nurses will be able to customize the web-based disease-specific instructions with the research team's help. They will reference these instructions as they perform discharge counseling and will give parents a copy of the instructions to refer to at home.
  Interventions: Other: Health Literacy-Informed Discharge Instructions
- Provider (Other): Baseline measures will be assessed for providers. They will then take part in a 20-minute training session, including information about health literacy, advanced counseling strategies, results of prior studies, and pre-implementation data. At the end of the study, assessments will be performed for those who use the health literacy-informed tool at least once during the study period.
  Interventions: Other: Provider Training

INTERVENTIONS:
Other: Health Literacy-Informed Discharge Instructions — Web-based disease-specific instruction sheets that will be printed with the research team's help. Providers will reference these instructions as they perform discharge counseling and will give parents a copy of the instructions to refer to at home.
  Arms: Parent: Post-Implementation
Other: Provider Training — 20-minute long provider training session, including information about health literacy, advanced counseling strategies, results of prior studies, and pre-implementation data.
  Arms: Provider

SUMMARY:
The overarching goal of this work is to identify strategies to reduce preventable pediatric post-hospitalization morbidity. In this study, investigators seek to address gaps in the knowledge base related to pediatric post-hospitalization morbidity by examining the understanding and execution of post-hospitalization discharge instructions in the context of low health literacy (HL).

DETAILED DESCRIPTION:
In this study, investigators seek to address gaps in the knowledge base related to pediatric post-hospitalization morbidity in 3 phases: first (Phase A) by examining the understanding and execution of post-hospitalization discharge instructions in the context of low HL, second (Phase B) by beginning to develop a low literacy discharge plan template to enhance and standardize provider counseling, and third (Phase C) by examining the effects of the intervention. The focus will be on those at greatest risk for low HL and poor outcomes, families from low SES backgrounds. Investigators therefore propose a prospective study (Phase A) to:

AIM 1. Examine associations between HL and parent execution of inpatient discharge instructions (overall and 4 key domains: medication management, follow-up, diet/activity restrictions, and concerning symptoms to act on;.

Hypothesis: Low HL will be adversely associated with execution (overall/individual domains).

AIM 2. Examine the role of understanding in the relationship between HL and parent execution of inpatient discharge instructions. a) Examine associations between HL and understanding (overall and 4 key domains). b) Examine the degree to which understanding mediates the relationship between HL and execution (overall and individual domains).

Hypothesis: Low HL will be adversely associated with understanding and its individual domains. The relationship between HL and execution will be partially mediated by understanding.

AIM 3 (Exploratory). Explore the role and mechanism through which low HL is related to post-hospitalization morbidity (as defined by readmissions, ED use, or unplanned doctor visits) by examining a) the association between HL and post-hospitalization morbidity, and b) the degree to which the relationship between HL and post-hospitalization morbidity occurs through overall understanding and execution.

Preliminary data from Phase A showed that >80% of parents make ≥1 error related to hospital discharge instructions. Notably, 30% of parents made medication errors, 20% missed >1 follow-up appointment, and 70% were not aware of concerning symptoms that should prompt medical attention. Findings from Phase A will be used to inform development of (Phase B) and to examine the efficacy of (Phase C) interventions to reduce post-hospitalization morbidity through a HL-informed approach as recommended by the Institute of Medicine. This work will build on a longstanding program of research and intervention development in this area by the study team.

The specific aims for Phases B and C are to:

AIM 4. Design a health literacy-informed discharge plan template tool to address domains of medication management, follow-up appointments, concerning symptoms to act on, and diet/activity restrictions.

AIM 5. Explore the efficacy of the tool in improving parent understanding and execution of discharge instructions (e.g. medication errors, appointment attendance, actions related to concerning symptoms, diet/activity restrictions).

Hypothesis: Parents will demonstrate improved understanding/execution of discharge instructions.

AIM 6. Explore the feasibility and utility of the tool with providers and parents.

Hypothesis: Providers/parents will find the tool to be easy to use and helpful.

ELIGIBILITY:
Parent

Inclusion Criteria:

* Primary caregiver of child ≤12 years old
* Primary caregiver of child discharged on ≥1 daily medication
* Primarily speaks and reads English or Spanish (by report).

Exclusion Criteria:

* Parent of child not discharged home (e.g. transferred to another facility<18 years old
* Vision difficulty (<20/50 corrected; Rosenbaum screener)
* Self-reported parent hearing difficulty

Provider

Inclusion Criteria:

* Pediatric resident at NYU School of Medicine

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 264 (Actual)
Dates: Start 2019-07-16 (Actual); Primary Completion 2020-03-12 (Actual); Study Completion 2020-04-02 (Actual)

PRIMARY OUTCOMES:
Parent Execution of Discharge Instructions | 14 days
  Execution will be assessed at three time points. The first assessment (T2) will take place in person, within the first two weeks of discharge, to coincide with a follow-up appointment if possible or at another convenient time for the parent. At this time point, execution will be assessed via structured survey and b) observed dosing assessment. Surveys will include information about execution of instructions related to medications (dose and adherence), follow up appointments (attendance), concerning symptoms, and restrictions. The electronic health record will also be reviewed to determine if appointments were attended

SECONDARY OUTCOMES:
Parent Understanding of Discharge Instructions | 1 day (within 12 hours of hospital discharge)
  Understanding will be measured in person or by phone after discharge education by the inpatient team but before parents begin administering scheduled home medications (T1b). Parents will be administered a structured survey. Actual understanding of medications, follow-up appointments, diet and activity restrictions, and concerning symptoms to monitor will be assessed. Questions will also include parent self-perceived understanding (including self-perceived understanding of medications, follow-up appointments, time of, diet and activity restrictions, and concerning symptoms). Subjects will rate their agreement with these statements on a 5 Point Likert Scale (Strongly Disagree to Strongly Agree). The adult version of this questionnaire has been validated and was later adapted for pediatric parents; we further modified this tool to include additional topics and to make it more easily understandable for parents with low literacy.
Post-Hospitalization Morbidity | 45 days
  Unplanned 7 and 30-day post-discharge readmissions, ED visits, and doctor visits) will be assessed via parent survey and via chart review.
Provider Outcomes: Baseline | Baseline: Day 1
  Survey at enrollment: Assessments include provider knowledge/attitudes/practices relating to counseling at the time of hospital discharge (assessment instrument modified from survey used in previous research study performed by this team).
Provider Outcomes | 45 days
  Follow-up survey: Providers who used the health-literacy informed tool at least once will be interviewed at the end of the study. Assessments include provider knowledge/attitudes/practices as well as perceived ease of use, utility, and barriers to use of the low literacy web-based intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Glick, MD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices). Requests should be directed to alexander.glick@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data.